CLINICAL TRIAL: NCT05483335
Title: Assessing the Frequency of Burnout Syndrome Among Medical Students in United Arab Emirates University and Identifying Any Associated Factors
Brief Title: Assessing Burnout in Medical Students in Clerkship Years in United Arab Emirates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Other Study IDs: UAEU_CMHS_IM_ERSC_2022_846
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Burnout, Student; Burnout, Professional; Educational Problems
Keywords: Medical Student; Clerkship; Burnout syndrome; Medical Education; Untied Arab Emirates
MeSH Terms: conditions — Burnout, Psychological; Burnout, Professional

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Student in the final two clinical years (Clerkship years): All the current medical students of College of Medicine and Health Sciences in United Arab Emirates University in the clinical years (fifth and sixth years in a 6-year MD programme) also called as clerkship years, will be invited into this study to assess for burnout syndrome using a validated tool via Mind GardenTM using Malasch Inventory for Burnout Syndrome and also to identify any other factors which may be contributing to stress/burnout.
  Interventions: Other: No intervention but assessing for burnout syndrome in all group

INTERVENTIONS:
Other: No intervention but assessing for burnout syndrome in all group — Using Maslach Burnout inventory to assess the presence of burnout and a self reporting questionnaire to identify possible stressors or associations

SUMMARY:
Burnout Syndrome is a medical condition caused by long-term job-related strain and is defined by presence of either one or more of the three states i.e. emotional exhaustion, depersonalization and lack of personal accomplishment. Burnout has been shown to cause decreased work output and mental well being of employees and increase errors at workplace. Burnout is observed in various lines of work and but has been found to be especially high among academic students undertaking professional studies as well as healthcare professionals. Medical students in their clerkship years undergo high stake exams, while adapting from classroom and simulation learning to participate in clinical care of patients in hospital care setting with no prior experience, which much them vulnerable to developing burnout during medical school. Burnout can effect medical students' well-being, which may continue into their internship and residency so greater emphasis in required on creating an awareness of burnout and identifying any factors associated to its development.

DETAILED DESCRIPTION:
Burnout syndrome can develop after a prolonged response to chronic emotional and interpersonal workplace stressors, and is defined by 3 dimensions - emotional exhaustion, depersonalization and lack of personal accomplishment. Burnout syndrome can be prevalent in up to half the medical students and those studies have suggested poor mental health among them. Various external and internal factors may contribute to burnout in medical students and little is known about the impact and mechanism of these factors in developing burnout. Burnout can develop, persist or worsen in residency years and it has been found to frequent among Diabetes specialty residents in United Kingdom as well in Emirati medical residents. Burnout can affect overall wellbeing of medical students with health consequences as well as poor work engagement/ educational outcomes.

To the best of authors knowledge no data exists on burnout in undergraduate medical students in clinical years (clerkship) in United Arab Emirates

ELIGIBILITY:
Inclusion Criteria:

1. Medical students (5th and 6th year) of college of medicine and health sciences in United Arab Emirates University
2. Currently attending the college, not on sick leave or long-term absence.
3. Agreed to participate after Informed consent

Exclusion Criteria:

Self-reported presence of active mental health illness or current treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Medical student of the 5th and 6th year (clinical/clerkship years) of the 6-year MD programme
  We plan to include at least 132 medical students based on sample size calculation with total population of 200 clerkship students with 95% confidence level and 5% margin of error.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assess the frequency of burnout syndrome in clerkship medical students (5th and 6th year of MD program) collected over 3 months period. | cross-sectional with data collected over 3 months
  The purpose of this study is to estimate the frequency of burnout syndrome in medical students in the clinical years (fifth and sixth years in a 6-year MD programme) in College of Medicine and Health Sciences in United Arab Emirates University via validated tool from Mind Garden, Malasch Inventory for Burnout Syndrome, assessing all three subscales of burnout i.e Emotional Exhaustion (with cutoff score for high burnout >26; range 0-54 with higher scores meaning a worse outcome), Depersonalization (with cutoff score for high burnout >12; range 0-30 with higher scores meaning a worse outcome), and lack of personal accomplishment (with cutoff score for high burnout < 32; range 0-48 with higher scores meaning a better outcome)
Assess factors associated with presence of burnout syndrome in clerkship medical students (5th and 6th year of MD program) collected over 3 months period. | cross-sectional with data collected over 3 months
  To identify factors associated with presence of burnout in medical students in the clinical years (fifth and sixth years in a 6-year MD programme) in College of Medicine and Health Sciences in United Arab Emirates University

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, Principal Investigator — United Arab Emirates University, College of Medicine & Health Sciences
Locations (1):
- Internal Medicine, College of Medicine and Health Sciences, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data with similar population for analysis in future

REFERENCES:
- [Background] Dyrbye LN, Thomas MR, Huntington JL, Lawson KL, Novotny PJ, Sloan JA, Shanafelt TD. Personal life events and medical student burnout: a multicenter study. Acad Med. 2006 Apr;81(4):374-84. doi: 10.1097/00001888-200604000-00010. PMID 16565189
- [Background] Ishak W, Nikravesh R, Lederer S, Perry R, Ogunyemi D, Bernstein C. Burnout in medical students: a systematic review. Clin Teach. 2013 Aug;10(4):242-5. doi: 10.1111/tct.12014. PMID 23834570
- [Background] Agha A, Basu A, Hanif W. Burnout in diabetes and endocrinology specialist registrars across England, Scotland and Wales in the pre-COVID era. Prim Care Diabetes. 2022 Aug;16(4):515-518. doi: 10.1016/j.pcd.2022.05.005. Epub 2022 Jun 3. PMID 35667990
- See also: The gold standard for burnout assessment. Maslach Burnout Inventory 4th Edition — http://www.mindgarden.com/117-maslach-burnout-inventory-mbi